CLINICAL TRIAL: NCT00003370
Title: A Trial of MGI 114 in Children With Solid Tumors: A Pediatric Oncology Group Phase I Cooperative Agreement Study
Brief Title: Irofulven in Treating Children With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01838; POG-9772; CDR0000066359 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2006-05

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — irofulven

ARMS (1):
- Arm I (Experimental): If the dose limiting toxicity is myelosuppression in stratum 1, then stratum 1 is closed and stratum 2 opens.
  Stratum 2 consists of the following: patients receiving no more than 2 prior chemotherapy regimens; patients who have not received prior central axis radiation or bone marrow transplantation; and patients with no known bone marrow involvement. Patients receive intravenous 6-hydroxymethylacylfulvene over 10 minutes daily for 5 days. The course is repeated every 28 days unless disease progression or unacceptable toxic effects are observed. Patients with stable or responding disease may receive up to 1 year of therapy. If dose limiting toxicity occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the maximum tolerated dose. Dose escalation will not occur until all patients within a cohort have been observed for 28 days from day 1 of therapy. Patients are followed until death.
  Interventions: Drug: irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
Phase I trial to study the effectiveness of irofulven in treating children with recurrent or refractory solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and dose limiting toxicity of 6-hydroxymethylacylfulvene (MGI-114) in pediatric patients with recurrent or refractory solid tumors.

II. Determine the incidence and severity of other toxic effects of MGI-114. III. Determine a safe and tolerable dose of MGI-114 to be used in phase II studies.

IV. Determine the pharmacokinetics of MGI-114 in these patients. V. Determine preliminary evidence of antitumor activity of MGI-114 against recurrent or refractory pediatric solid tumors.

OUTLINE: This is a dose escalation study. If the dose limiting toxicity is myelosuppression in stratum 1, then stratum 1 is closed and stratum 2 opens.

Stratum 2 consists of the following: patients receiving no more than 2 prior chemotherapy regimens; patients who have not received prior central axis radiation or bone marrow transplantation; and patients with no known bone marrow involvement. Patients receive intravenous 6-hydroxymethylacylfulvene over 10 minutes daily for 5 days. The course is repeated every 28 days unless disease progression or unacceptable toxic effects are observed. Patients with stable or responding disease may receive up to 1 year of therapy. If dose limiting toxicity occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the maximum tolerated dose. Dose escalation will not occur until all patients within a cohort have been observed for 28 days from day 1 of therapy. Patients are followed until death.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven recurrent or refractory solid tumors
* No leukemia
* Patients with brain tumors are not eligible until the first 2 patients at each dose level are evaluable for toxicity

PATIENT CHARACTERISTICS:

* Age: 21 and under
* Performance status: Karnofsky 50-100% Lansky play scale 50-100% (for infants)
* Life expectancy: At least 8 weeks
* Absolute neutrophil count at least 1,000/mm3
* Hemoglobin at least 9 g/dL
* Platelet count at least 75,000/mm3
* Bilirubin less than 1.5 mg/dL
* SGPT less than 5 times upper limit of normal
* Creatinine normal for age OR GFR at least 70 mL/min
* Cardiac shortening fraction at least 27% OR institutional normal OR cardiac ejection fraction greater than 50% OR institutional normal
* Neurologic deficits in patients with CNS tumors must be stable for at least 2 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after the study
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

* At least 1 week since prior growth factor therapy and recovered
* At least 6 months since prior bone marrow transplantation and no evidence of graft versus host disease
* At least 2 weeks since prior myelosuppressive chemotherapy and recovered
* At least 6 weeks since prior nitrosourea and recovered
* At least 2 weeks on stable dexamethasone for patients with CNS tumors
* No concurrent chemotherapy
* At least 2 weeks since prior palliative radiotherapy (small port)
* At least 6 months since prior substantial bone marrow radiation
* At least 6 months since total abdominal, pelvic, chest, mantle, and Y ports radiotherapy
* No other concurrent anticancer therapy or investigational agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 1998-08; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail C. Megason, MD, Study Chair — University of Mississippi Cancer Clinic
Locations (56):
- United States (51):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Veterans Affairs Medical Center - Huntington, Huntington, West Virginia
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Bomgaars LR, Megason GC, Pullen J, Langevin AM, Dale Weitman S, Hershon L, Kuhn JG, Bernstein M, Blaney SM. Phase I trial of irofulven (MGI 114) in pediatric patients with solid tumors. Pediatr Blood Cancer. 2006 Aug;47(2):163-8. doi: 10.1002/pbc.20686. PMID 16317728